CLINICAL TRIAL: NCT04765163
Title: Research on Intelligent Assist System of Colonoscope Operating Handle
Brief Title: Research on Operating Handle of Colonoscope
Acronym: ROHC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XXT17
Record Dates: First submitted 2021-01-26; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Colonic Disease
Keywords: Intelligence; Colonocope; Handle
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- physician group with assistive equipment: The number of colonoscopy operations completed per unit time and the degree of fatigue in the physician group using assistive equipment
  Interventions: Device: Intelligent Operating Handle
- Physician group without assistive equipment: The number of colonoscopy operations completed per unit time and the degree of fatigue in the physician group without assistive equipment

INTERVENTIONS:
Device: Intelligent Operating Handle — Intelligent Operating Handle
  Groups: physician group with assistive equipment

SUMMARY:
Artificial intelligence is deeply integrated with medical diagnosis, and intelligent colonoscopy technology has broad room for development. At present, the assist device of colonoscopy is insufficiently studied. It is the part that needs to be further explored in the development of artificial intelligence colon diagnosis and treatment technology. The study will be conducted at the Digestive Endoscopy Center and it is expected that 380 subjects will participate voluntarily. Subjects met: 1) routine colonoscopy; 2) willing to provide relevant information required by the experiment; 3) signed informed consent for the study. This topic focuses on the colonoscope assist device, through the combination of power assisting device, dynamic analysis, and migration expert skills, to achieve a combination of intelligent power and precise treatment, and establish a prototype of the patient-colonoscopy-assisted assist system-doctor's four-in-one diagnosis and treatment system.

ELIGIBILITY:
Inclusion Criteria:

1. routine colonoscopy;
2. Willing to provide relevant information required by this experiment;
3. Sign the informed consent form for this study.

Exclusion Criteria:

1. can not tolerate colonoscopy;
2. Information about the requirements of this study cannot be provided;
3. Questionnaires cannot be conducted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: After full informed consent, outpatients undergoing a physical examination for colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2019-05-11 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Colonoscope operating handle model | January 21, 2021
  CPAS-I/II prototype system

SECONDARY OUTCOMES:
Patents | November 11, 2020
  1. Patent number: 202010389077.8, A non-slip sleeve and a colonoscope handle
  2. Patent number: 202010388602.4, A colonoscopy operation auxiliary glove
  3. Patent number: 202011112968.5, A colonoscope control device

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Ruigang, Beijing, China